CLINICAL TRIAL: NCT03329859
Title: Impact of Microcomplications in Laparoscopic Surgery on Operative Time and Costs - Multimodal Strategy to Reduce Microcomplications
Brief Title: Microcomplications in Lap. Cholecystectomy: Reducing Intraoperative Interruptions by High Resolution Standardization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: EK10/12
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Workflow; Costs; Laparoscopy; Cholecystectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): "High resolution standardized laparoscopic cholecystectomy" Patients in which laparoscopic cholecystectomy was performed after high Resolution standardization and Training of the OR Team according to the Standard.
  Interventions: Procedure: High resolution standardized laparoscopic cholecystectomy
- Control arm (Active Comparator): No 'High resolution standardized laparoscopic cholecystectomy' Patients in which laparoscopic cholecystectomy was performed in the conventional way without prior standardization
  Interventions: Procedure: High resolution standardized laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: High resolution standardized laparoscopic cholecystectomy — High resolution standardized laparoscopic cholecystectomy

SUMMARY:
Objective: Investigators aimed to evaluate the impact of a high resolution standardized laparoscopic (HRSL) cholecystectomy protocol on operative time and intraoperative interruptions in a teaching hospital.

Background: Interruptions of the surgical workflow or microcomplications (MC) lead to prolonged procedure times and costs and can be indicative for surgical mistakes. Reducing MC can improve operating room efficiency and prevent intraoperative complications.

Methods: Audio video records of laparoscopic cholecystectomies were reviewed regarding type, frequency and duration of MC before and after the implementation of a HRSL which included the introduction of a stepwise protocol for the procedure and a teaching video. After consent operating team members were obliged to prepare the operation with these resources.

ELIGIBILITY:
Inclusion Criteria:

* age above and including 18 years
* indication for laparoscopic cholecystectomy
* written informed consent of patient
* written informed consent of the operating team

Exclusion Criteria:

* age below 18 years
* other laparoscopic or open surgical procedure in the same operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
median hourly delay due to microcomplications | Any microcomplications are recorded between skin incision to skin closure during laparoscopic cholecysectomy
  median hourly increase in operative time in seconds due to microcomplications before and after an intervention to reduce microcomplications. Microcomplications are defined as any interruption of the surgical workflow.

CONTACTS AND LOCATIONS:
Overall Officials: Marco von Strauss und Torney, MD, Principal Investigator — University Hospital Basel, Department of General and Visceral Surgery, Spitalstrasse 21, CH-4031 Basel
Locations (1):
- University Hospital Basel/Dep. of General and Visceral Surgery, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] von Strauss Und Torney M, Aghlmandi S, Zeindler J, Nowakowski D, Nebiker CA, Kettelhack C, Rosenthal R, Droeser RA, Soysal SD, Hoffmann H, Mechera R. High-resolution standardization reduces delay due to workflow disruptions in laparoscopic cholecystectomy. Surg Endosc. 2018 Dec;32(12):4763-4771. doi: 10.1007/s00464-018-6224-y. Epub 2018 May 21. PMID 29785458